CLINICAL TRIAL: NCT06858800
Title: Pinch Grip and Functional Outcomes betweenHematoma Distraction Arthroplasty Versus Ligament Reconstruction Tendon Interposition Arthroplasty in Trapeziometacarpal Osteoarthritis: A Randomized Clinical Trial
Brief Title: Pinch Grip and Functional Outcomes Between Hematoma Distraction Arthroplasty Versus Ligament Reconstruction Tendon Interposition Arthroplasty in Trapeziometacarpal Osteoarthritis.
Acronym: Rhizarthrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de la Santa creu i Sant Pau - Barcelona (Other)
Collaborators: Universitat Autonoma de Barcelona (Other); Hospital de Mollet (Unknown)
Responsible Party: Principal Investigator, Anna Castellà Pujol, Resident of Orthopaedics and Traumatology, Hospital de la Santa creu i Sant Pau - Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIC-20161003
Record Dates: First submitted 2025-02-04; First posted 2025-03-05 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis Thumbs; Rhizarthrosis; Trapeziometacarpal (TMC) Arthrosis
Keywords: Osteoarthritis; Thumb; Rhizarthrosis; Trapezectomy; Arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Before each intervention, the type of procedure to perform was determined using a balanced simple randomization computer system to allocate treatments provided by the surgical area supervisor to the surgeon in the operation room.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ligament reconstruction with tendon interposition (LRTI) technique (Experimental): A complete removal of the trapezium bone through a radial-volar incision was performed, with a subsequent resection of the posterior articular surface of the first metacarpal bone. A ligament transfer using a loop from a hemi-tendonectomy of the flexor carpi radialis (FCR) was used to cushion the joint and occupy the space left by the resected bone, following the modified Weilby-Garcia-Elias technique.
  Interventions: Procedure: LTRI technique
- Hematoma distraction Artroplasty (HDA) technique (Experimental): A dorso-radial incision in the CMC joint was used in order to perform a trapeziectomy. The thumb was repositioned to its anatomical position (subtle opposition with 30º abduction) and fixed percutaneously with a 1.5 mm K-wire for three weeks along with a cast. This allowed the postoperative hematoma to act as an interposition between the first metacarpal and the scaphoid.
  Interventions: Procedure: HDA technique

INTERVENTIONS:
Procedure: LTRI technique — Hematoma distraction Artroplasty (HDA): A dorso-radial incision in the CMC joint was used in order to perform a trapezectomy. The thumb was displaced at its anatomical position (subtle opposition with 30º abduction) and fixed percutaneously with a 1.5mm K-Wire for three weeks along with a cast. This allowed to act the postoperative hematoma as an interposition between first-metacarpal and the scaphoid.
  Ligament reconstruction with tendon interposition (LRTI): A complete removal of the trapezium bone with a radial-volar incision was made with posterior resection of the articular surface of the first metacarpal bone, and ligament transfer with a loop from hemi-tendonectomy of the flexor carpi radialis (FCR) was used to cushion the joint while occupying the space of the resected bone following modified Weilby Garcia-Elias technique
  Arms: Ligament reconstruction with tendon interposition (LRTI) technique
Procedure: HDA technique — A dorso-radial incision in the CMC joint was used in order to perform a trapezectomy. The thumb was displaced at its anatomical position (subtle opposition with 30º abduction) and fixed percutaneously with a 1.5mm K-Wire for three weeks along with a cast. This allowed to act the postoperative hematoma as an interposition between first-metacarpal and the scaphoid
  Other Names: Hematoma distraction Artroplasty
  Arms: Hematoma distraction Artroplasty (HDA) technique

SUMMARY:
To date, there is no gold standard for the treatment of severe trapeziometacarpal joint osteoarthritis. Despite the fact that new procedures have been described, techniques such hematoma distraction or ligament reconstruction tendon interposition are still valid non-implant options. The main hypothesis was that patients treated with LTRI technique would show superior clinical outcomes at one-year follow-up in terms of tip and key pinch and DASH scores in comparison with HDA technique. As secondary objectives, complication rates and surgical times were recorded.

ELIGIBILITY:
Inclusion Criteria:

Patients who attended the hand unit's outpatient clinic at a regional trauma center with a diagnosis of grade III-IV TMC OA according to the Eaton-Littler radiological scale, who had previously failed conservative treatments (NSAIDs, splints, RHB, and corticosteroid injections) and desired surgical intervention with sufficient comprehension to participate in this study.

Exclusion Criteria:

Previous procedures on the same extremity distal to the elbow, central or peripheral neurological disease, and patient withdrawal.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Functional results between HDA and LTRI using the QuickDASH test | From enrollment to end of follow-up at 1 year
  Functional results were collected preoperatively and at 12 months postoperatively at the same facility, with a one-year follow-up. The score used to measure function and symptoms was the QuickDASH questionnaire. Patients responded to 11 statements, rating them from 1 to 5. Scores ranged from 0 (no disability) to 100 (most severe disability). Clinical evaluation and data collection were performed by a level 2 specialist, according to Tang et al.'s criteria of the Hand Unit.
Clinical results between HDA and LTRI with the quantification of grip and tip pinch strenght with JAMAR dynanometer. | From enrollment to end of follow-up at 1 year
  Grip and tip pinch strength were quantified using a BASELINE® hydraulic pinch gauge and dynamometer. Each patient completed three maximal pinch attempts, and the highest value was used for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Creu i Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Maybe we will share IDP used in the results publications